CLINICAL TRIAL: NCT06911372
Title: The Impact of Gestational Diabetes Mellitus on Cerebral Blood Flow and Cerebrovascular Function After Pregnancy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Anna Stanhewicz, PhD (Other)
Responsible Party: Sponsor-Investigator, Anna Stanhewicz, PhD, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 202410260
Record Dates: First submitted 2025-03-12; First posted 2025-04-04 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Gestational Diabetes Mellitus (GDM); Postpartum Women; Uncomplicated Pregnancy
Keywords: Gestational Diabetes; Brain Blood Flow; Pregnancy; Postpartum
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vascular Tests (Experimental): All women will complete the same protocol, regardless of pregnancy history.
  Interventions: Drug: Intradermal Microdialysis; Other: Brain Blood Flow Tests; Other: Local Heating

INTERVENTIONS:
Drug: Intradermal Microdialysis — A total of three microdialysis sites will be perfused with ringer's solution, L-NAME, or ketorolac (one drug per site). After a baseline period, all three sites will undergo tests of blood vessel function including an acetylcholine dose-response protocol and a test of maximal skin blood flow with sodium nitroprusside.
Other: Brain Blood Flow Tests — Participants will complete CO2 breathing procedures to evaluate brain blood vessel health.
Other: Local Heating — A dime-sized heater will be placed on the skin to evaluate cutaneous microvascular function

SUMMARY:
Gestational Diabetes Mellitus (GDM) currently affects approximately 14% of all pregnancies worldwide. Importantly, the health-related consequences of GDM extend well beyond pregnancy, such that women with a history of GDM have a 40% increased risk of cerebrovascular diseases and a 67% increased risk of dementia, compared to women with a history of uncomplicated pregnancy. Women with a history of GDM have impaired skin microvascular function, compared with women with a history of uncomplicated pregnancy. Therefore, it's likely that GDM results in impaired brain blood vessel function, yet there is little-to-no information regarding the effects of GDM on brain blood vessel health and function after pregnancy.

Therefore, the purpose of the study is to evaluate the effects of GDM on brain blood flow and brain blood vessel function in healthy women with either a history of GDM or uncomplicated pregnancy.

In this study, the investigators will use two different types of ultrasound to non-invasively measure brain blood flow. Brain blood vessel function will be evaluated by examining the brain blood flow responses to increases in carbon dioxide (the increases in carbon dioxide are similar to what is experienced during a breath hold). Additionally, the investigators will compare the brain blood flow results to skin microvascular function to explore potential mechanisms behind possible impairments in brain blood vessel function. Skin microvascular function will be assessed using a minimally invasive technique (intradermal microdialysis for the local delivery of pharmaceutical agents) on dime sized areas of the forearm. Finally, for screening purposes and to further explore potential mechanisms behind any potential impairments in brain blood vessel function, the investigators will perform blood draws to determine the metabolic health of the participants and to analyze for substances that influence blood vessel function.

ELIGIBILITY:
INCLUSION CRITERIA:

* Post-partum women
* 18 years or older
* Delivered within 5 years from the study visit
* History of gestational diabetes diagnosed by an obstetrician and confirmed according to the American College of Obstetricians and Gynecologists criteria for gestational diabetes OR history of uncomplicated pregnancy (defined as no history of gestational diabetes, hypertensive pregnancy, or other gestational disorder).

EXCLUSION CRITERIA: We exclude participants from both groups for:

* Skin diseases
* Current tobacco use
* Diagnosed or suspected hepatic or metabolic disease including diabetes
* Diagnosed with depression or other mood-related disorders, asthma, chronic obstructive pulmonary disease, cystic fibrosis, or pulmonary fibrosis
* Use of prescribed NSAIDs, statins or other cholesterol-lowering medication, antihypertensive medication, carbonic anhydrase inhibitors, corticosteroids, thyroid medications, antidepressants or mood stabilizers, diuretics, phenothiazines, or benzodiazepines
* History of preeclampsia or gestational hypertension,
* History or family history of panic disorder,
* Currently pregnant
* Body mass index <18.5 kg/m2,
* Allergy to materials used during the experiment (e.g. latex), known allergies to study drugs.
* History of heavy alcohol use/binge drinking,
* Have planned procedures with radiological contrast,
* Have a major dental procedure/surgery coming up, such as a dental extraction
* Anatomy of the middle cerebral artery or internal carotid artery that prevents adequate ultrasonography and/or and data collection

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2028-04-15 (Estimated)

PRIMARY OUTCOMES:
Stepped hypercapnia-induced change in middle cerebral artery velocity | During the study visit, an average of 5 hours
  Middle cerebral artery velocity responses to stepped concentrations of inhaled carbon dioxide gas
Hypercapnia-induced change in internal carotid artery diameter | During the study visit, an average of 5 hours
  Internal carotid artery shear-mediated dilation response to inhaled carbon dioxide
Change in microvascular blood flow response to increasing concentrations of acetylcholine | During the study visit, an average of 5 hours
  Cutaneous vascular vasodilator responses to acetylcholine perfusion in lactated Ringer's, ketorolac, and L-NAME treated microdialysis sites.

CONTACTS AND LOCATIONS:
Locations (1):
- Iowa Bioscience Innovation Facility, Iowa City, Iowa, United States